CLINICAL TRIAL: NCT03958942
Title: Effect of Bilateral Ultrasound Guided Quadratus Lumborum Block Versus Lumbar Epidural Block on Postoperative Analgesia, and Inflammatory Response Following Major Lower Abdominal Cancer Surgery
Brief Title: Bilateral Ultrasound Guided Quadratus Lumborum Versus Lumbar Epidural Block on Postoperative Analgesia, and Inflammatory Response in Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, assisstant professor of Anesthesia, ICU, and Pain Management, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 255
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain; Inflammatory Response
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- quadratus lumborum block (Active Comparator): received pre-emptive ultrasound-guided quadratus lumborum block with 25 mL of 0.25% bupivacaine on each side of the abdominal wall before induction of GA.
  Interventions: Other: Ultrasound quadratus lumborum block with bupivacaine 25%
- lumbar epideural block (Active Comparator): received pre-emptive lumbar epidural block with 15 mL of 0.25% bupivacaine before induction of GA.
  Interventions: Other: lumbar epideural block with bupivacaine 25%

INTERVENTIONS:
Other: Ultrasound quadratus lumborum block with bupivacaine 25% — echogenic needle will be inserted in-plane with the ultrasound beam in a posterior-to-anterior direction through the quadratus lumborum muscle until the ventral fascia of the muscle penetrated. At this point, the needle directed toward the fascial plan between the quadratus lumborum and the Psoas muscle
  Arms: quadratus lumborum block
Other: lumbar epideural block with bupivacaine 25% — lumbar epidural will be performed for patients in group II using a 16-gauge Touhy epidural needle by a median approach. The T12 - L1 or L1 - L2 interspaces will be chosen for the injection. The epidural space identified by the loss of resistance technique.
  Arms: lumbar epideural block

SUMMARY:
This study aims at comparing the effects of bilateral ultrasound-guided quadratus lumborum block versus lumbar epidural block on postoperative analgesia and inflammatory response following major lower abdominal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA II, III
* Weight 50 - 85 kg.
* Scheduled for major lower abdominal cancer surgery (radical cystectomy, total abdominal hysterectomy).

Exclusion Criteria:

* Patients with a history of relevant drug allergy.
* Coagulation disorders.
* Opioid dependence.
* Sepsis.
* Local infection at the vicinity of the block site.
* Patients with psychiatric illnesses that would interfere with perception and assessment of pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | first 24 hours postoperatively
  postoperative pain intensity.

SECONDARY OUTCOMES:
postoperative inflammatory response | first 24 hours postoperatively
  inflammatory response represented by the levels of: interleukins 1,6, and tumor necrosis factor alpha
side effects | first 24 hours postoperatively
  sedation, nausea, vomiting, and respiratory depression

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided